CLINICAL TRIAL: NCT06949683
Title: Effects of Meal and Exercise Sequence on Glucose and Blood Pressure Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202310HM014-1
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Glucose Response; Blood Pressure
Keywords: Fasted-exercise; Post-Exercise Hypotension; Postprandial glucose responses; Blood pressure
MeSH Terms: conditions — Post-Exercise Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal-Exercise (Experimental): Breakfast intake before 22 minutes of brisk walking
  Interventions: Behavioral: Meal-Exercise
- Exercise-Meal (Experimental): 22 minutes of brisk walking before breakfast intake
  Interventions: Behavioral: Exercise-Meal

INTERVENTIONS:
Behavioral: Meal-Exercise — Breakfast intake before 22 minutes of brisk walking, followed by a lunch intake for another 75 minutes of observation period. The entire experiment lasted a total of 150 minutes.
  Arms: Meal-Exercise
Behavioral: Exercise-Meal — 22 minutes of brisk walking before breakfast intake, followed by 75 minutes of observational period. The entire experiment lasted a total of 150 minutes
  Arms: Exercise-Meal

SUMMARY:
The purpose of this study is to investigate whether the sequence meal and exercise (exercise before meal or exercise after meal) affects the postprandial metabolism.

DETAILED DESCRIPTION:
Trial days In the 24 h prior to each main trial, participants were asked to refrain from performing any strenuous physical activity and from consuming alcohol/caffeine. Dinner intake was recorded before the first main trial and participants were asked to replicate this diet prior to their second main trial.

On main trial days, participants arrived at the laboratory between 8-9 am following a 10-hour fast. After measuring height, blood pressure, pulse, and obtaining finger-prick blood samples, participants underwent EM or ME intervention.

The entire experiment lasted a total of 150 minutes. During the initial 50 minutes, participants were randomly assigned to either exercise before or after breakfast. Participants were asked to finish their breakfast within approximately 5 minutes. The exercise regimen consisted of brisk walking for 22 minutes at a speed of 6 km/hr on the indoor track. After a 25-minute break, the second meal was provided. Participants then underwent a 75-minute observation period during the postprandial phase. Blood pressure and pulse were assessed with the individual seated in a relaxed, upright position on a chair, with the arm properly positioned. Two measurements of blood pressure and pulse were taken, and these values were averaged to ensure that the two readings were within 5 mmHg of each other. If the two readings differed by more than 5 mmHg, additional readings were taken until the outlying measurement was excluded. The test meal consists of red bean dorayaki (CHUAN LIAN Enterprise Co., Ltd.) and soy milk (I-MEI Foods Co., Ltd.). The breakfast provided contained 348 kcal, with a macronutrient distribution of 60% carbohydrates, 12% protein, and 28% fat. The second meal contained 207 kcal, with a macronutrient distribution of 66% carbohydrates, 6% protein, and 28% fat.

Finger-prick blood samples, blood pressure, and pulse were measured every 25 minutes during the experiment using the Freestyle Optium Neo (Abbott Diabetes Care, Ltd., UK) and the OMRON HEM-7320 blood pressure monitor (OMRON Co., Ltd., Japan). Two measurements of blood pressure and pulse were taken, and these values were averaged to ensure that the two readings were within 5 mmHg of each other. If the two readings differed by more than 5 mmHg, additional readings were taken until the outlying measurement was excluded. Blood pressure and pulse were assessed with the individual seated in a relaxed, upright position on a chair, with the arm properly positioned.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 45 years
2. Body Mass Index (BMI) ranging from 18.5 to 27 kg/m2
3. No habits of heavy drinking or smoking, or have quit smoking for at least 6 months
4. Absence of diabetes, cardiovascular, or metabolic-related disorders
5. Not currently taking medications, or other supplements that may affect blood sugar, blood pressure, or metabolic changes
6. No current sports injuries or medical advice against exercise
7. No significant weight fluctuations in the past three months (within ±3% of usual body weight)
8. Not experiencing shift work or travel across time zones within the past 6 months
9. No current plans to change lifestyle habits and willing to adhere to the requirements of the study

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose concentrations | 150 minutes
  Changes in glucose responses during trials
Blood pressure | 150 minutes
  Changes in blood pressure (e.g., diastolic and systolic blood pressure) during trials

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan